CLINICAL TRIAL: NCT05335356
Title: A Randomized, Double-Blind, Parallel Group, Multicenter, Phase 3 Study to Compare the Efficacy and Safety of Bmab 1200 and Stelara in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Comparing Efficacy and Safety of Bmab 1200 and Stelara in Patients With Moderate to Severe Chronic Plaque Psoriasis
Acronym: STELLAR-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocon Biologics UK Ltd (Industry)
Responsible Party: Sponsor
Organization: Biocon Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM12H-PSO-03-G-02
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blinded (Patient, Investigator),
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bmab1200 (Experimental): Bmab 1200 45 mg Bmab 1200 90 mg
  Interventions: Biological: Bmab1200
- Stelara (Active Comparator): Stelara 45 mg Stelara 90 mg
  Interventions: Biological: Stelara

INTERVENTIONS:
Biological: Stelara — 45 mg , 90 mg at Week 0, 4, 16, 28 and 40;During the study after receiving 2 doses , before dosing at Week 16 patients were re-randomised in a 1:1 ratio to receive either Bmab 1200 or Stelara .
  Arms: Stelara
Biological: Bmab1200 — 45 mg , 90 mg at Week 0, 4, 16, 28 and 40
  Arms: Bmab1200

SUMMARY:
This is a randomized, double-blind, active-controlled, parallel-group, multicenter study designed to compare the efficacy, safety, immunogenicity, and PK(Pharmacokinetic) of Bmab 1200 with Stelara in adult patients with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
Approximately 384 patients with moderate to severe plaque psoriasis will be enrolled and randomly assigned to one of the 2 treatment groups in a 1:1 ratio (192 patients in the Bmab 1200 group and 192 patients in the Stelara group). Patients who are diagnosed as moderate to severe chronic plaque psoriasis for at least 6 months and are candidate for systemic therapy or phototherapy at the time of the screening visit will be enrolled. The study is planned to be conducted in Europe and North America across approximately 48 sites in 5 countries. The study will be conducted in an outpatient setting, and the participation for each patient will consist of a screening period (up to 4 weeks/28 days) and a double-blind, active-controlled treatment period (52 weeks) with a rerandomization step for switching therapy (Bmab 1200 with Stelara ) before Week 16 dosing. The treatment period before the switch is TP1(Treatment Period1) and post switch is TP2(Treatment Period 2) (from Week 16 dosing to prior to Week 28 dosing) and TP3 (Treatment Period3)(from Week 28 dosing to Week 52). The total duration of the study (excluding the screening period) will be 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide informed consent form (ICF), able to follow study instructions, and comply with the protocol requirements as per the investigator's opinion.
2. Patient is aged 18 to 80 years, both inclusive, and weighing <130 kg at the time of the screening visit.
3. Patient has a diagnosis of chronic plaque psoriasis for at least 6 months and is a candidate for systemic therapy or phototherapy at the time of the screening visit.
4. Patient with moderate to severe chronic plaque psoriasis as defined by BSA (Body surface area)involvement

   * 10%, PASI score ≥12, and sPGA ≥3 at the screening and baseline visits.
5. Patient has stable disease for at least 2 months before the baseline visit (ie, without clinically significant changes in the investigator's opinion).
6. Patient has adequate renal and hepatic function at the screening
7. Women of childbearing potential must have a negative serum pregnancy test during screening and a negative urine pregnancy test at baseline. A female patient is considered not of childbearing potential when postmenopausal or surgically sterilized
8. Women of childbearing potential and male patients with a female partner of childbearing potential must be willing to use highly effective contraceptive precautions.

Exclusion Criteria:

1. Patient has nonplaque psoriasis, such as erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, other skin conditions (eg, eczema), other current or chronic systemic autoimmune or inflammatory disease at the time of screening visit that would interfere with the evaluation of the effect of the study treatment on psoriasis. Patients with concurrent psoriatic arthritis will be allowed to participate.
2. Patient who has a current or past history of any of the following infections:

   1. Current or past history of congenital or acquired immunodeficiency or patient is positive for the human immunodeficiency virus (HIV) antibodies (HIV-1 or HIV-2) at screening.
   2. Patient has current infection with hepatitis B virus (HBV) or hepatitis C virus (HCV) as per serological tests at screening.

      * For HBV, patients who test positive to hepatitis B surface antigen (HBsAg) will be excluded. Patients who test positive to hepatitis B core antibody (HBcAb) only (HBsAg negative), may be enrolled if they also test positive to hepatitis B surface antibody (HBsAb).
      * For HCV, patient who test positive to HCV antibody will be excluded unless they test negative for HCV RNA.
   3. Presence of active infection at screening or history of infection requiring intravenous antibiotics and/or hospitalization ≤8 weeks before baseline visit, or oral/intramuscular antibiotics ≤4 weeks before baseline visit, or topical antibiotics ≤2 weeks before baseline visit. Minor localized fungal infections or topical antibiotics for facial acne may be allowed.
   4. Any recurrent bacterial, fungal, opportunistic or viral infection including recurrent/disseminated herpes zoster that, based on the investigator´s clinical assessment, causes a safety risk and makes the patient unsuitable for the study.
   5. History of invasive/systemic fungal infection (eg, histoplasmosis) or nontubercular mycobacterial infection.
3. Patient meeting any of the following tuberculosis (TB)-related conditions:

   1. Patient who has current or history of active TB.
   2. Patient who has signs or symptoms suggestive of active TB upon medical history or physical examination including chest radiography at screening. If a chest radiography performed within the past 3 months before screening is available, it does not need to be repeated at screening.
   3. Patients with current latent TB (defined as a positive result of interferon-γ release assay [IGRA] with a negative examination of chest radiography [posterior-anterior and lateral views, or per country regulations where applicable] and absence of symptoms). Patients with positive IGRA (Interferon Gamma Release Assay) may be enrolled if they have documentation of completed appropriate country-specific TB prophylaxis within the past 5 years or have received at least 1 month of country-specific TB prophylaxis before the baseline visit and are willing to complete its entire course, and do not have other risk factors, radiologic findings, or physical evidence supporting latent or active TB. If a patient's initial IGRA test result is indeterminate, the test can be repeated once. If the test result is again indeterminate, the patient will be excluded from the study.
   4. Patient who has had exposure to a person with active TB, such as first-degree family members or coworkers within 16 weeks before the baseline visit.
4. Patient has an underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic including central nervous system demyelinating disease, endocrine, cardiac, infection, or gastrointestinal) which, in the opinion of the investigator, significantly immune-compromises the patient and/or places the patient at unacceptable risk for receiving an immunomodulatory therapy.
5. Patient had a major surgical intervention within 12 weeks of the baseline or planned major surgery during the study period.
6. Patient who has prior exposure to more than 1 biologic agent for the treatment of psoriasis or psoriatic arthritis.
7. Patient who has received or plans to receive any of the prohibited medications or treatment that could affect psoriasis:
8. Patient has received a live or live-attenuated vaccine within 4 weeks before the baseline visit. Patient must agree not to receive a live or live-attenuated vaccine during the study and up to 15 weeks after the last dose of the study treatment.
9. Patient who has had Bacillus Calmette-Guérin (BCG) vaccination within 1 year before the baseline visit. Patients must agree not to receive a BCG vaccination during the study and at least 1 year after the last dose of the study treatment.
10. Have a transplanted organ/tissue or stem cell transplantation.
11. TP3 specific criteria:

    1. Patient is willing and able to provide revised informed consent form (ICF), able to follow study instructions, and comply with the protocol requirements as per the investigator's opinion
    2. Patient has not developed any condition/ or met study discontinuation or treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Apex Clinical Research Center, Mayfield Heights, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szepietowski JC, Reich A, Feldman SR, Pulka G, Mekokishvili L, Tsiskarishvili N, Svarca I, Poder A, Singh G, Deodhar S, Kumar K, Marwah A, Loganathan S, Wolff-Holz E, Athalye SN. Comparative efficacy and safety of biosimilar Bmab 1200 versus reference ustekinumab in moderate-to-severe plaque psoriasis: 52-week findings from the Phase 3 STELLAR-2 trial. Expert Opin Biol Ther. 2025 Oct;25(10):1121-1133. doi: 10.1080/14712598.2025.2576506. Epub 2025 Oct 21. PMID 41100115
- [Derived] Szepietowski JC, Reich A, Feldman SR, Pulka G, Mekokishvili L, Tsiskarishvili N, Svarca I, Poder A, Singh G, Deodhar S, Kumar K, Marwah A, Loganathan S, Athalye SN, Wolff-Holz E. Efficacy and safety of the ustekinumab biosimilar, Bmab 1200, versus reference ustekinumab in moderate-to-severe plaque psoriasis: 28-week results of the randomized, double-blind, Phase 3 STELLAR-2 study. Expert Opin Biol Ther. 2025 Aug;25(8):913-924. doi: 10.1080/14712598.2025.2538608. Epub 2025 Jul 29. PMID 40708530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Europe and North America and enrolled patients across 41 sites in 5 countries.
Groups:
- Bmab1200; Stelara: Eligible patients were randomly assigned in a 1:1 ratio to receive Bmab 1200 or Stelara based on predefined stratification factors of geographic region (US vs Europe), body weight (≤100 kg vs >100 kg), previous exposure to biologic-based therapies (Yes vs No), and concomitant psoriatic arthritis (Yes vs No). Patients received study treatment at the baseline visit and Week 4. Patients weighing ≤100 kg received a subcutaneous dose of 45 mg of either drug at each of the above visits, while patients weighing >100 kg received a subcutaneous dose of 90 mg (45 mg × 2).
- Bmab 1200- Bmab 1200; Stelara-Stelara; Stelara-Bmab 1200: Before dosing at Week 16, patients in the Stelara group were randomly assigned in a 1:1 ratio to receive either Bmab 1200. This was done to obtain data after a single switch in patients who had been treated with Stelara.
  All continuing patients who received study treatment with Bmab 1200 at the baseline visit and Week 4 and achieved at least PASI 50 response by Week 12 were rerandomized before receiving study treatment at Week 16. This was done to maintain the study blinding, i.e. the patients in the original Bmab 1200 group went through the rerandomization procedure; however, they were assigned and continued to receive Bmab 1200.
- Bmab 1200/Bmab 1200; Stelara/Stelara; Stelara/Bmab 1200: All continuing patients who completed TP2 (received study treatment at the baseline visit and Weeks 4 and 16) and achieved at least PASI 75 response at Week 28 were offered to enter TP3 of the study to continue the same treatment that they were rerandomized to receive during TP2 (Bmab 1200 or Stelara) in a blinded manner. For patients not eligible to enter TP3, the end of study (EOS) visit occurred at Week 28.
Period: Treatment Period 1 (Baseline to Week 16)
Arm/Group | Bmab1200 | Stelara | Bmab 1200- Bmab 1200 | Stelara-Stelara | Stelara-Bmab 1200 | Bmab 1200/Bmab 1200 | Stelara/Stelara | Stelara/Bmab 1200
Started | 191 | 193 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 190 | 192 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Week 16 to Week 28)
Arm/Group | Bmab1200 | Stelara | Bmab 1200- Bmab 1200 | Stelara-Stelara | Stelara-Bmab 1200 | Bmab 1200/Bmab 1200 | Stelara/Stelara | Stelara/Bmab 1200
Started | 0 | 0 | 185 | 94 | 92 | 0 | 0 | 0
Completed | 0 | 0 | 171 | 87 | 86 | 0 | 0 | 0
Not Completed | 0 | 0 | 14 | 7 | 6 | 0 | 0 | 0
Period: Treatment Period 3 (Week 28 to Week 52)
Arm/Group | Bmab1200 | Stelara | Bmab 1200- Bmab 1200 | Stelara-Stelara | Stelara-Bmab 1200 | Bmab 1200/Bmab 1200 | Stelara/Stelara | Stelara/Bmab 1200
Started | 0 | 0 | 0 | 0 | 0 | 168 | 81 | 84
Completed | 0 | 0 | 0 | 0 | 0 | 163 | 79 | 82
Not Completed | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patient demographics and baseline characteristics provided on FAS which consist of all participants who signed the ICF and were randomized
Groups:
- Stelara: Stelara 45 mg Stelara 90 mg
  Stelara: 45 mg , 90 mg at Week 0, 4, 16, 28 and 40; Before dosing at Week 16, patients in the Stelara group were randomly assigned in a 1:1 ratio to receive either Bmab 1200 or Stelara
- Total: Total of all reporting groups
Arm/Group | Bmab1200 | Stelara | Total
Number analyzed (Participants) | 191 | 193 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.09) | 43.9 (13.58) | 43.2 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 57 | 127
  Male | 121 | 136 | 257
Race/Ethnicity, Customized [Number; unit: Subject]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 185 | 187 | 372
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 190 | 192 | 382
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: Subject]
  Europe | 189 | 189 | 378
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Psoriasis Area and Severity Index (PASI)
Description: Percentage change from baseline in the Psoriasis Area and Severity Index score at Week 12
Time Frame: Baseline to Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | Bmab1200 | Stelara
Number analyzed (Participants) | 191 | 193
Percentage change from baseline | -79.87 (2.818) | -80.55 (2.783)

2. Secondary Outcome: PASI Score
Description: Percentage change from baseline in the PASI score at Baseline through Week 28.
  PASI is a quantitative rating score for measuring the severity of psoriatic lesions based on area coverage, plaque appearance, their response to therapy. 4 regions- head, upper limbs, trunk, and lower limbs are assessed separately for erythema, induration/thickness, and scaling. Degree of involvement is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement) for each region. Total score (sum of erythema, thickness, and scaling) is multiplied by the degree of involvement for each body region and then multiplied by constant. Sum of all lesion scores can range from 0 (no disease) to 72 (maximal disease), with the higher score indicating more severe disease. Change from baseline in PASI score indicates response to therapy. PASI 50 means ≥50% reduction from baseline in the PASI score
Time Frame: Baseline through Week 28
Measure: Mean (Standard Deviation); unit: Percentage change from Baseline in Score
Groups:
- Stelara-Bmab 1200: Bmab 1200 45 mg 90 mg Stelara 45 mg 90 mg
  Subject who received Stelara 45 mg dose have received Bmab 1200 dose 45 mg Subject who received Stelara 90 mg dose have received Bmab 1200 dose 90 mg
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 168 | 81 | 84
Percentage change from Baseline in Score | -95.50 (6.068) | -96.01 (6.461) | -95.44 (7.321)

3. Secondary Outcome: PASI Improvement
Description: PASI improvement of ≥50% relative to baseline (PASI 50), PASI improvement of ≥75% relative to baseline (PASI 75), and PASI improvement of ≥90% relative to Baseline through Week 28 and 52
  PASI is a quantitative rating score for measuring the severity of psoriatic lesions based on area coverage, plaque appearance, their response to therapy. 4 regions- head, upper limbs, trunk, and lower limbs are assessed separately for erythema, induration/thickness, and scaling. Degree of involvement is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement) for each region. Total score (sum of erythema, thickness, and scaling) is multiplied by the degree of involvement for each body region and then multiplied by constant. Sum of all lesion scores can range from 0 (no disease) to 72 (maximal disease), with the higher score indicating more severe disease. Change from baseline in PASI score indicates response to therapy. PASI 50 means ≥50% reduction from baseline in the PASI score
Time Frame: Baseline through Week 28
Measure: Count of Participants; unit: Participants
Groups:
- Stelara-Stelara: Before dosing at Week 16, patients in the Stelara group were randomly assigned in a 1:1 ratio to receive either Bmab 1200 or Stelara Those patients who were randomized to Stelara received a further 2 doses as given below Stelara 45 mg, patients weighing <100 kg at Week 16, and 28 ; Stelara 90 mg, patients weighing >100 kg at Week 16, and 28 ;
- Stelara-Bmab 1200: Those patients who were receiving stelara and randomised to Bmab1200 received a further 1 dose in TP3 as given below Bmab 1200 45 mg, patients weighing <100 kg at Week 40 ; Bmab 1200 90 mg, patients weighing >100 kg at week 40
Arm/Group | Bmab1200 | Stelara-Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 168 | 80 | 84
Participants
  PASI 50 | 168 | 80 | 84
  PASI 75 | 168 | 79 | 83
  PASI 90 | 140 | 70 | 67

4. Secondary Outcome: Static Physician's Global Assessment (sPGA)
Description: Change from Baseline in sPGA During TP2.
  The sPGA is a quantitative rating score of the patient's psoriasis based on physician's assessment at a given time point according to the following categories: induration, erythema, and scaling. The sPGA is a 6-point scale and patient's psoriasis is graded as clear (0), minimal (1), mild (2), moderate (3), marked (4), severe (5). The sum of the scores for induration, erythema, and scaling will be divided by 3 to obtain a final sPGA score. lower score indicates better disease status
Time Frame: Baseline through Week 28
Population: sPGA-(averaged over all lesions); Score range: 0-5 Induration (I): 0 (no plaque-elevation) to 5 (severe plaque-elevation); Erythema (E): 0 (no erythema, hyperpigmentation maybe present) to 5 (dusky to deep-red coloration); Scaling (S): 0 (no scaling) to 5 (severe-very thick tenacious scale) sPGA based on Total-Average (I+E+S= /3): 0 (Cleared, except for residual discoloration) to 5 (Severe, majority of lesions have individual scores for I+E+S/3 that averages 5) Refer Apndx3-Protocol V3.0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 168 | 81 | 84
score on a scale | -3.0 (1.21) | -2.9 (1.21) | -2.8 (1.28)

5. Secondary Outcome: Affected Body Surface Area
Description: Change from baseline in affected body surface area at Weeks 28
  Total % BSA afflicted by psoriasis is estimated using a handprint of the patient at each visit . The entire palmar surface of the patient's handprint is assumed to correspond to approximately 1% of total BSA. Reduction in BSA indicates improvement
Time Frame: Baseline through Week 28
Measure: Mean (Standard Deviation); unit: Percentage of total body surface area
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 168 | 81 | 84
Percentage of total body surface area | -26.52 (15.152) | -25.91 (13.323) | -28.33 (17.251)

6. Secondary Outcome: Dermatology Life Quality Index Scores
Description: Change from baseline in quality of life as measured by Dermatology Life Quality Index scores at Weeks 28
  It is a 10-item patient-reported outcome questionnaire that, in addition to evaluating overall QoL, can be used to assess 6 different aspects that may affect QoL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Nine of the 10 questions have response categories including "not relevant" (score of 0), "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3); Question 7 is a "yes"/ "no" question where "yes" is scored as 3. Eight items also have a "Not relevant" option scored "0," which indicates no problems. Total scores range from 0 to 30 (less to more impairment) and a 5-point change from baseline is considered a clinically important difference.
Time Frame: Baseline through Week 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 170 | 90 | 88
score on a scale | -12.2 (6.84) | -10.5 (6.74) | -12.2 (7.08)

7. Secondary Outcome: Dermatology Life Quality Index Scores
Description: Change from baseline in quality of life as measured by Dermatology Life Quality Index scores at Weeks 52
  It is a 10-item patient-reported outcome questionnaire that, in addition to evaluating overall QoL, can be used to assess 6 different aspects that may affect QoL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Nine of the 10 questions have response categories including "not relevant" (score of 0), "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3); Question 7 is a "yes"/ "no" question where "yes" is scored as 3. Eight items also have a "Not relevant" option scored "0," which indicates no problems. Total scores range from 0 to 30 (less to more impairment) and a 5-point change from baseline is considered a clinically important difference.
Time Frame: Baseline through Week 52
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 152 | 79 | 79
score on a scale | -12.8 (6.73) | -11.5 (6.35) | -12.7 (6.98)

8. Secondary Outcome: Static Physician's Global Assessment (sPGA)
Description: Change in Static Physician's Global Assessment (sPGA) at Weeks 52
  The sPGA is a quantitative rating score of the patient's psoriasis based on physician's assessment at a given time point according to the following categories: induration, erythema, and scaling. The sPGA is a 6-point scale and patient's psoriasis is graded as clear (0), minimal (1), mild (2), moderate (3), marked (4), severe (5). The sum of the scores for induration, erythema, and scaling will be divided by 3 to obtain a final sPGA score. lower score indicates better disease status
Time Frame: Baseline through Week 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 163 | 80 | 82
score on a scale | -3.1 (1.21) | -3.0 (1.29) | -2.9 (1.20)

9. Secondary Outcome: Affected Body Surface Area
Description: Change from baseline in affected body surface area at Weeks 52
  Total % BSA afflicted by psoriasis is estimated using a handprint of the patient at each visit . The entire palmar surface of the patient's handprint is assumed to correspond to approximately 1% of total BSA. Reduction in BSA indicates improvement
Time Frame: Baseline through Week 52
Measure: Mean (Standard Deviation); unit: Change from Baseline in %BSA
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 163 | 80 | 83
Change from Baseline in %BSA | -27.42 (15.119) | -26.50 (13.160) | -28.90 (17.560)

10. Secondary Outcome: PASI Improvement
Description: PASI improvement of ≥50% relative to baseline (PASI 50), PASI improvement of ≥75% relative to baseline (PASI 75), and PASI improvement of ≥90% relative to Week 52
Time Frame: Baseline through week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 163 | 80 | 83
Participants
  PASI 50 | 163 | 80 | 83
  PASI 75 | 159 | 80 | 81
  PASI 90 | 133 | 70 | 63

11. Other Pre Specified Outcome: Safety:-Treatment-emergent Adverse Events Including Adverse Events of Special Interest and Adverse Reactions During the Treatment Period
Time Frame: Baseline to Week 52
Measure: Count of Participants; unit: Participants
Groups:
- Stelara-Bmab1200: Bmab 1200 45 mg 90 mg Stelara 45 mg 90 mg
  Subject who received Stelara 45 mg dose have received Bmab 1200 dose 45 mg Subject who received Stelara 90 mg dose have received Bmab 1200 dose 90 mg
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab1200
Number analyzed (Participants) | 191 | 101 | 92
Participants
  Endometrial adenocarcinoma | 1 | 0 | 0
  Squamous cell carcinoma of the tongue | 1 | 0 | 0
  Angioedema | 0 | 1 | 0
  Rash maculo-papular | 0 | 1 | 0
  Abdominal pain | 1 | 0 | 0
  Jaundice cholestatic | 1 | 0 | 0
  Alcohol poisoning | 0 | 1 | 0

12. Other Pre Specified Outcome: Safety:- Injection-site Reactions
Description: Injection-site reactions at Day 1, Week 4, Week 16, and throughout the study
Time Frame: Baseline through Week 28 and 52
Population: NAb status with no injection site reactions being reported.
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab1200
Number analyzed (Participants) | 0 | 0 | 0

13. Other Pre Specified Outcome: Safety:- Hypersensitivity
Description: Hypersensitivity at Day 1, Week 4, Week 16, and throughout the study
Time Frame: Baseline through Week 52
Measure: Number; unit: participants
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 191 | 101 | 92
participants | 1 | 3 | 1

14. Other Pre Specified Outcome: Immunogenicity:-Developing Antidrug Antibodies
Description: Proportion of patients developing antidrug antibodies
Time Frame: Baseline through Week 28
Population: n = number of patients with available data
Measure: Number; unit: participants
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 185 | 94 | 92
participants
  ADA positive | 162 | 88 | 86
  ADA negative | 21 | 6 | 5
  Patients with no post baseline ADA result | 2 | 0 | 1

15. Other Pre Specified Outcome: Immunogenicity:-Developing Antidrug Antibodies
Description: Proportion of patients developing antidrug antibodies
Time Frame: Postdosing Week 52
Population: n = number of patients with available data
Measure: Number; unit: participants
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 168 | 81 | 84
participants
  ADA positive | 131 | 73 | 74
  ADA negative | 36 | 8 | 10
  Patients with no post baseline ADA result | 1 | 0 | 0

16. Other Pre Specified Outcome: Developing Neutralizing Antibodies
Description: Proportion of patients neutralizing antibodies
Time Frame: Baseline through Week 28
Population: n = number of patients with available data
Measure: Number; unit: participants
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 162 | 88 | 86
participants
  Nab reactive | 54 | 42 | 31
  Nab negative | 108 | 46 | 55

17. Other Pre Specified Outcome: Developing Neutralizing Antibodies
Description: Proportion of patients neutralizing antibodies
Time Frame: Postdosing Week 52
Population: n = number of patients with available data
Measure: Number; unit: participants
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 131 | 73 | 74
participants
  Nab reactive | 27 | 19 | 12
  Nab negative | 104 | 54 | 62

18. Other Pre Specified Outcome: Pharmacokinetic:-Serum Concentrations
Description: Serum concentrations of ustekinumab
Time Frame: Postdosing on Week 28
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Bmab 1200 (1 Injection); Stelara-Stelara (1 Injection); Stelara-Bmab 1200 (1 Injection): Patients who weigh ≤100 kg: Stelara® 45 mg (1 injection of 45 mg PFS)
- Bmab 1200 (2 Injection); Stelara-Stelara (2 Injection); Stelara-Bmab 1200 ((2 Injection): Patients who weigh >100 kg: Stelara® 90 mg (2 injections of 45 mg PFS)
Arm/Group | Bmab 1200 (1 Injection) | Stelara-Stelara (1 Injection) | Stelara-Bmab 1200 (1 Injection) | Bmab 1200 (2 Injection) | Stelara-Stelara (2 Injection) | Stelara-Bmab 1200 ((2 Injection)
Number analyzed (Participants) | 130 | 61 | 61 | 36 | 15 | 20
ng/mL | 678.308 (444.7791) | 589.780 (418.9308) | 620.793 (398.1352) | 796.833 (392.6448) | 1070.600 (522.0039) | 861.665 (549.4014)

19. Other Pre Specified Outcome: Pharmacokinetic:-Serum Concentrations
Description: Serum concentrations of Ustekinumab
Time Frame: Postdosing on Week 52
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Stelara-Bmab 1200 (2 Injection): Patients who weigh >100 kg: Stelara® 90 mg (2 injections of 45 mg PFS)
Arm/Group | Bmab 1200 (1 Injection) | Stelara-Stelara (1 Injection) | Stelara-Bmab 1200 (1 Injection) | Bmab 1200 (2 Injection) | Stelara-Stelara (2 Injection) | Stelara-Bmab 1200 (2 Injection)
Number analyzed (Participants) | 127 | 60 | 61 | 35 | 17 | 20
ng/mL | 728.029 (477.1775) | 665.403 (379.9506) | 653.908 (415.8309) | 881.343 (510.0086) | 1008.382 (671.8667) | 898.450 (551.4494)

20. Secondary Outcome: PASI Score
Description: Percentage change from baseline in the PASI score at Baseline through Week 52.
  The PASI (Psoriasis Area and Severity Index) is a score from 0 to 72 that measures psoriasis severity based on lesion redness, thickness, scaling, and body area affected. The body is divided into four regions, each scored separately. Scores are calculated using severity and area involvement, and are used to assess treatment response (e.g., PASI 50 = 50% improvement).
Time Frame: Baseline through Week 52
Measure: Mean (Standard Deviation); unit: Percentage change from Baseline
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab 1200
Number analyzed (Participants) | 163 | 81 | 84
Percentage change from Baseline | -95.50 (7.507) | -96.60 (5.671) | -94.71 (7.950)

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events (TEAEs) through the Study (Week 52)
Arm/Group | Bmab1200 | Stelara | Stelara-Bmab1200
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/101 | 0/92
Serious Adverse Events (participants affected / at risk) | 6/191 | 0/101 | 1/92
Other Adverse Events (participants affected / at risk) | 111/191 | 48/101 | 51/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bmab1200 (N=191) | Stelara (N=101) | Stelara-Bmab1200 (N=92)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bmab1200 (N=191) | Stelara (N=101) | Stelara-Bmab1200 (N=92)
Nasopharyngitis (Infections and infestations) | 18 (23) | 6 (6) | 8 (8)
Influenza (Infections and infestations) | 4 (4) | 5 (8) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 1 (1) | 6 (7)
Urinary tract infection (Infections and infestations) | 6 (6) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 4 (4) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (2)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tongue fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 12 (14) | 6 (9) | 2 (3)
Blood triglycerides increased (Investigations) | 11 (13) | 3 (4) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 6 (7) | 2 (2) | 1 (1)
Blood cholesterol increased (Investigations) | 4 (6) | 2 (3) | 2 (2)
Blood pressure increased (Investigations) | 3 (3) | 2 (2) | 2 (2)
Blood glucose increased (Investigations) | 2 (3) | 3 (3) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Weight increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Lipids increased (Investigations) | 1 (1) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Acquired mixed hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Latent autoimmune diabetes in adults (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Erythropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Secondary thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 3 (3)
Leukocyturia (Renal and urinary disorders) | 3 (3) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Ketonuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperoxaluria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 0 (0)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (2) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Illness anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data are the property of the Sponsor and cannot be published without prior authorization from the Sponsor, but data and publication thereof will not be unduly withheld.

DOCUMENTS (2):
  • Study Protocol (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT05335356/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT05335356/SAP_001.pdf